CLINICAL TRIAL: NCT02482649
Title: Equine-Assisted Activities and Therapy for Treating Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: EAA/Therapy for Treating Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-12-049
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics; Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EAA/T (Experimental): EAA/TEquine-Assisted Activities and Therapy) bi-weekly for 12eeks
  Interventions: Behavioral: EAA/T
- Drugs (Active Comparator): Methylphenidate or Atomoxetine
  Interventions: Drug: Methylphenidate; Drug: Atomoxetine

INTERVENTIONS:
Behavioral: EAA/T — bi-weekly for 12weeks
  Other Names: Equine-Assisted Activities and Therapy; Hyppotherapy
  Arms: EAA/T
Drug: Methylphenidate — dosage adjustment according to clinical effectiveness, QD for 12weeks
  Other Names: Cencerta; Metadate
  Arms: Drugs
Drug: Atomoxetine — dosage adjustment according to clinical effectiveness, QD or BID, for 12weeks
  Other Names: Strattera
  Arms: Drugs

SUMMARY:
The aim of this study is 1) to investigate clinical effects of equine-assisted activities and therapy (EAA/T) for treating attention-deficit/hyperactivity disorder (ADHD) and 2) to compare the clinical effect of EAA/T and drug therapy in children 6-13-years-of-age. This study is designed as a 12-week, prospective, open labeled trial, including 24 sessions of EAA/T. Forty six subjects will be enrolled and various clinical tests will be administered at baseline and after EAA/T or drug therapy.

DETAILED DESCRIPTION:
This study is designed as a 12-week, prospective, open labeled trial, including 24 sessions of EAA/T. Forty six subjects will be aasigned 12 weeks of EAA/T or drug therapy, and various clinical tests will be administered at baseline and after EAA/T or drug therapy. Assessments included the investigator-administered ADHD-Rating Scale (ARS-I), Clinical Global Impressions - Severity scale (CGI-S), Clinical Global Impressions - Improvement scale (CGI-I), Gordon Diagnostic System (GDS), Korea-Child Behavior Checklist (K-CBCL), Self-Esteem Scale (SES), Bruininks-Oseretsky test of motor proficiency, second edition (BOT-2), and quantitative electroencephalography (QEEG) or functional magnetic resonance imaging(fMRI) study. This study has two objectives. The first objective is to investigate clinical effects of equine-assisted activities and therapy (EAA/T) for treating attention-deficit/hyperactivity disorder (ADHD). For this one, we determine the treatment response rate as the primary outcome measure. The treatment response is defined as ≥ 30% decline than baseline in the ARS-I score or in CGI-I scores of 1 or 2 to endpoint. The second objective is to compare the clinical effect of EAA/T and drug therapy in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of ADHD according to Diagnostic and Statistical Manual-IV-Text Version(DSM-IV-TR) and Korean Kiddie-Schedule for Affective Disorders and Schizophrenia-Present and Life¬time Version (K-SADS-PL)

Exclusion Criteria:

* (1) a learning disorder or an intelligence quotient (IQ) measured by the Korean Wechsler Intelligence Scale for Children-IV (K-WISC-IV) < 70, (2) significant medical condition, schizophrenia or other psychotic disorder, bipolar disorder, a history of alcohol or drug dependence, neurologic disorders, epilepsy, and organic mental disorders; (3) a major depressive disorder that required pharmacotherapy; (4) significant suicidal ideation; (5) a Tourette's disorder or obsessive-compulsive disorder that required pharmacotherapy; (6) use of methylphenidate or atomoxetine within 90 days of baseline

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
chane of ARS-I score | change measures (baseline and 12 weeks)
  change of Investigator-administered ADHD-Rating Scale (ARS-I) after Equine-Assisted Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Sook Joung, M.D.,Ph.D., Principal Investigator — Department of Psychiatry, Samsung Medical Center
Locations (1):
- Yoo-Sook Joung, Seoul, South Korea